CLINICAL TRIAL: NCT00231244
Title: Sirolimus-Eluting BX VELOCITYTM Balloon-Expandable Stent in a Compassionate Use Registry
Brief Title: Sirolimus-Eluting BX VELOCITYTM Balloon-Expandable Stent in a Compassionate Use Registry (SECURE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sid Cohen, MD, Cordis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P01-6310
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): CYPHER Sirolimus-Eluting Coronary Stent
  Interventions: Device: CYPHER Sirolimus-Eluting Coronary Stent

INTERVENTIONS:
Device: CYPHER Sirolimus-Eluting Coronary Stent — CYPHER Sirolimus-Eluting Coronary Stent

SUMMARY:
The objective of this study is to allow treatment with the sirolimus-eluting Bx VELOCITYTM stent in patients with a serious disease or condition for which there is no generally acceptable alternate treatment available.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female patient minimum 18 years of age
2. There is no alternative treatment for this patient as determined by the treating physician and an uninvolved cardiac surgeon;
3. Target lesion is 2.50mm and 3.50mm in diameter (visual estimate);
4. Target lesion is 45mm in length (visual estimate), treated with a maximum of three 18 mm stents;

Exclusion Criteria:

1. There is currently another method of treatment for the patient, including coronary artery bypass surgery (CABG) or brachytherapy;
2. The study target lesion has definite or possible thrombus present by angiographic criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2002-03; Primary Completion 2008-05 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is a composite of Target Vessel Failure (TVF) defined as target vessel revascularization, myocardial infarction or cardiac death at 30 days, 6mo, 12mo, 2, 3, 4, and 5 years. | 30 days, 6mo, 12mo, 2, 3, 4, and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Teirstein, MD, Principal Investigator — Scripps Clinic and Research
Locations (1):
- Scripps Clinic and Research, La Jolla, California, United States

REFERENCES:
- [Background] Costa M, Angiolillo DJ, Teirstein P, Gilmore P, Leon M, Moses J, Yakubov S, Carter A, Fischell T, Zenni M, Bass T. Sirolimus-eluting stents for treatment of complex bypass graft disease: insights from the SECURE registry. J Invasive Cardiol. 2005 Aug;17(8):396-8. PMID 16079441